CLINICAL TRIAL: NCT05500157
Title: Assessment of Treatment With Laparoscopic Fenestration or Aspiration Sclerotherapy for Large Symptomatic Hepatic Cysts (ATLAS): a Randomized Clinical Trial.
Brief Title: Assessment of Treatment With Laparoscopic Fenestration or Aspiration Sclerotherapy for Large Symptomatic Hepatic Cysts
Acronym: ATLAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-7134
Record Dates: First submitted 2022-05-06; First posted 2022-08-12 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-05

CONDITIONS: Liver Cyst; Polycystic Liver Disease; Autosomal Dominant Polycystic Kidney; Autosomal Dominant Polycystic Liver Disease
Keywords: polycystic liver disease; aspiration sclerotherapy; fenestration
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration sclerotherapy (Active Comparator): Aspiration sclerotherapy is a percutaneous procedure that evacuates fluid from the liver cyst and subsequently exposes cyst lining to a sclerosing agent (e.g. ethanol, minocycline) for a limited period of time.
  Interventions: Procedure: aspiration sclerotherapy versus laparoscopic fenestration
- Laparoscopic Fenestration (Active Comparator): Laparoscopic fenestration exposes the liver through laparoscopic surgery. During this procedure the cyst is punctured and drained followed by resection of the extra-hepatic cyst wall
  Interventions: Procedure: aspiration sclerotherapy versus laparoscopic fenestration

INTERVENTIONS:
Procedure: aspiration sclerotherapy versus laparoscopic fenestration — See arm description

SUMMARY:
Patients with large hepatic cysts (> 5cm) may develop symptoms. These can be captured with the polycystic liver disease questionnaire (PLD-Q). Treatment of large hepatic cysts consists of aspiration sclerotherapy or laparoscopic fenestration.

The safety and efficacy of both procedures has been explored in two recent systematic reviews yet no evident conclusion regarding superiority of either procedure could be drawn.

The main objective of the ATLAS trial is to compare laparoscopic fenestration and aspiration sclerotherapy in patients with large symptomatic hepatic cysts on patient-reported outcomes.

DETAILED DESCRIPTION:
Rationale: Patients with large hepatic cysts(>5cm) may develop symptoms due to distention of Glisson's capsule and/or compression on other abdominal organs. Frequently reported symptoms include abdominal pain, early satiety, nausea, and dyspnea. These symptoms can be captured in the disease-specific Polycystic Liver Disease Questionnaire (PLD-Q), a validated instrument. The treatment of symptomatic liver cysts is aimed to improve symptoms and quality of life by reducing cyst volume. There are two procedures available to treat symptomatic liver cysts: percutaneous aspiration sclerotherapy and laparoscopic fenestration.

In aspiration sclerotherapy, fluid is evacuated from the liver cyst and subsequently the cyst lining is exposed to a sclerosing agent for a limited period of time. Sclerotherapy causes temporary recurrence of cyst fluid after drainage, but subsequently results in a steady decrease of cyst volume in the majority of patients.

In laparoscopic fenestration the liver is exposed through laparoscopic surgery. In this procedure the cyst is punctured and drained followed by resection of extra-hepatic cyst wall.

The safety and efficacy of aspiration sclerotherapy and laparoscopic fenestration have been explored in two recent systematic reviews. No evident conclusion could be drawn because of the retrospective study design in the vast majority of the studies and the heterogeneity among these. A randomized controlled trial is warranted to identify the possible differences in safety and efficacy in aspiration sclerotherapy and laparoscopic fenestration.

Hypothesis: The investigators expect patients treated with laparoscopic fenestration to have better clinical outcome; i.e. a lower PLD-Q score, compared to aspiration sclerotherapy, when measured 4 weeks after the procedure. The investigators expect this difference to become smaller over time (after 6 and 12 months), with loss of statistical significance.

Objective: The main objective is to compare laparoscopic fenestration and aspiration sclerotherapy in patients with large symptomatic hepatic cysts on patient-reported outcomes. This information can be used to assess cost-effectiveness in both treatments.

Study design: A prospective, randomized clinical superiority trial in which patients will be randomized 1:1 to one of the treatment arms. Patients will be followed for 1 year.

Study population: All patients ≥18 years who are diagnosed with a dominant, simple hepatic cyst (>5 cm in diameter), that are symptomatic (PLD-Q score ≥20) and have an indication for treatment (both aspiration sclerotherapy and laparoscopic fenestration) are suitable for inclusion in this study. Only patients that are eligible for both treatments can be included in this study. In particular, patients with multiple cysts (>20 cysts of >1.5 cm) will be excluded as surgery leads to more complications in these patients.

Intervention: Patients will be randomly allocated to either aspiration sclerotherapy or laparoscopic fenestration. Both procedures are performed according to the standard Radboudumc protocols. Aspiration sclerotherapy consists of ultrasound-guided, percutaneous drainage of the cyst with subsequent sclerosation with ethanol. Laparoscopic fenestration consists of standard abdominal laparoscopy in which the large cyst(s) are drained and deroofed.

Main study parameters: The main study parameter is the PLD-Q score at 4 weeks after treatment. Secondary parameters are among others: PLD-Q score at baseline, 6 months and 12 months; liver volume (CT) at baseline and 4 weeks; cyst volume (ultrasound) at baseline, 4 weeks, 6 months and 12 months; complications according to Clavien-Dindo; admission duration, recurrence and re-intervention rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hepatic cyst characteristics:

  * Large (>5 cm),
  * Symptomatic (PLD-Q score ≥20),
  * Non-parasitic on imaging (US/CT/MRI)
  * Non-neoplastic on imaging (US/CT/MRI)
* Providing informed consent

Exclusion Criteria:

* Clinical indication of a complicated hepatic cyst (cyst rupture or active cyst infection)
* Cyst is not laparoscopically accessible for surgery
* Cyst is not percutaneously (ultrasound-guided) accessible for aspiration
* More than 20 cysts of >1.5 cm
* Age above 75 years
* ASA IV
* ECOG score >1
* Aspiration sclerotherapy or laparoscopic fenestration of hepatic cysts was performed in the last 6 months.
* Severe renal impairment (eGFR < 30 ml/min/1,73 m2)
* Coagulopathy (spontaneous INR >2 or platelet count < 80 x 109/l)
* Radiologic contrast allergy
* Pregnancy
* Any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator (e.g. inability to fill out questionnaires).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
PLD-Q 4 weeks | 4 weeks after the procedure
  Comparison of PLD-Q scores 4 weeks after the procedure, adjusted for baseline PLD-Q score.

SECONDARY OUTCOMES:
PLD-Q score 1, 6 and 12 months after intervention | up to 12 months
  PLD-Q score at 1, 6 and 12 months after intervention, adjusted for baseline
PLD-Q invididual symptoms | up to 12 months
  PLD-Q individual symptom scores at 1, 6 and 12 months after intervention, compared to baseline
SF-36 MCS | up to 12 months
  SF-36 Mental Component Score at 1, 6 and 12 months after intervention, adjusted to baseline
SF 36 PCS | up to 12 months
  SF-36 Physical Component Score at 1, 6 and 12 months after intervention, adjusted to baseline
EQ-5D-5L | up to 12 months
  EQ-5D-5L score at 1, 6 and 12 months after intervention, adjusted to baseline
Liver and cyst volume | up to 12 months
  Liver and cyst volume with CT before and 12 months after the intervention
Liver and cyst volume at recurrence | up to 12 months
  Liver and cyst volume in cases of recurrence of symptoms
Cyst volume with US | up to 12 months
  Cyst volume with ultrasound, at baseline and 1, 6 and 12 months after intervention.
Adverse events | up to 12 months
  Adverse events (according to Clavien-Dindo)
Technical success | periprocedural
  Technical success
Hospital stay | periprocedural
  Hospital stay in days
Re-intervention rates | up to 12 months
  Re-intervention rates during 12 months follow-up.
Cost-effectiveness iPCQ | up to 12 months
  Cost-effectiveness of both procedures iPCQ 1, 6 and 12 months after intervention, adjusted for baseline
Cost-effectiveness iMCQ | up to 12 months
  Cost-effectiveness of both procedures iMCQ 1, 6 and 12 months after intervention, adjusted for baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joost P.H. Drenth, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available to other researchers for clinical research purposes upon reasonable request to the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will be provided upon reasonable request with the principal investigator
Access Criteria: Study data will be provided upon reasonable request with the principal investigator